CLINICAL TRIAL: NCT02483832
Title: Effects of Message Framing and Risk Feedback on CRC Screening
Brief Title: Message Framing and Colorectal Cancer Screening
Acronym: CRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00057568
Record Dates: First submitted 2015-06-25; First posted 2015-06-29 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gain-frame (Active Comparator): This group will receive messages about the benefits of colorectal cancer screening.
  Interventions: Behavioral: Educational materials
- Loss-frame (Active Comparator): This group will receive messages about the disadvantages of not getting colorectal cancer screening.
  Interventions: Behavioral: Educational materials

INTERVENTIONS:
Behavioral: Educational materials — Educational materials about colorectal cancer and how to get screened will be presented to participants, with either gain- or loss-frame messages associated.

SUMMARY:
The main purpose of this study is to promote colorectal cancer (CRC) screening among individuals who have never been screened, with these individuals being members of a panel who participant in online studies. The primary study goals are to test effects of the matching between level of comparative risk feedback for colorectal cancer (CDC), that is, how one's risk compares to others, and message framing (Gain vs. loss frame) on CRC screening intentions and screening as well as mediators of effects in the context of people who obtain CRC risk feedback and framing messages online (i.e., Internet).

DETAILED DESCRIPTION:
1. Purpose and objective: The investigators propose an online intervention to increase colorectal cancer screening among men and women ages 50 to 75 who have never been screened for this disease. The intervention consists of giving study participants information about their estimated risk of getting colorectal cancer followed by either a message emphasizing the benefits of getting screened (i.e., gain frame messages) or the disadvantages of not getting screened (loss frame messages). Before conducting the online intervention, the investigators will conduct a pilot study to validate the gain and loss frame messages.
2. Study activities and population group: The pilot study activities involve recruiting 20 participants, screening for eligibility and conducting informed consent over the phone, randomizing them to receive either gain or loss frame messages, and instructing them to complete a survey with questions covering comprehension and framing manipulation checks. Data entry and survey activities will all be conducted through a secure REDCap project.

   Main study activities involve a pilot conducted by GfK involving 40 participants, 20 randomized to gain and 20 to the loss conditions, completing an online baseline survey and a post-intervention online survey. In addition, participants are to review: 1) educational materials on colorectal cancer and colorectal cancer screening, 2) review and respond to questions about their estimated risk of getting colorectal cancer, and 3) review and respond to questions about gain- or loss-framed messages. After the pilot, the full study will begin. Study activities will be the same as in the pilot, with the addition of a six month post-intervention online survey.
3. Data analyses and risk/safety issues: Analyses will include descriptive statistics and use of linear and logistic regression analyses. Every effort will be made to ensure the confidentiality of the information collected. During the pilot study, the only PHI recorded is an email address for the purposes of conducting the online surveys, a physical address so that the study team can send a copy of the consent form, and information for payment. Demographic information and email address will be recorded during phone screening and entered into a secure REDCap database after the participant has given informed consent, and an internal record ID will be generated for the participant in REDCap that will be used to identify them throughout the study. Physical address and payment information will be recorded after informed consent. All paper data will be destroyed as soon as possible.

In the main study run by GfK, all data received by the key personnel from Gfk will be de-identified per GfK policy. There are no foreseeable physical risks; although some participants in the main study may be surprised by their risk estimate and react negatively (e.g., experience some anxiety) if the estimate is very high.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-75
* able to read and write English
* never had colorectal cancer
* never had colorectal cancer screening tests

Exclusion Criteria:

* History of colorectal cancer
* history of colorectal cancer screening tests

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 640 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2015-08-24 (Actual); Study Completion 2015-08-24 (Actual)

PRIMARY OUTCOMES:
CRC screening follow-up rate | Six months
  Respondents will be required to complete a six-month follow-up survey and answer questions about any CRC screening they have sought out and/or completed since the intervention.

SECONDARY OUTCOMES:
Changes in attitudes towards CRC and CRC screening as measured by survey | Baseline, immediately post-intervention, six months
  Respondents will be required to complete a baseline survey (with questions before the intervention and immediately after the intervention) and a six-month follow-up survey that includes the same questions on attitudes towards CRC and CRC screening. We will compare the results to assess changes in attitudes before intervention, immediately after intervention, and six months after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Lipkus, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University School of Nursing, Durham, North Carolina, United States